CLINICAL TRIAL: NCT01888445
Title: A Japanese, Phase 2, Multicenter, Randomized, 4-arm Parallel, Double-blind (Arms 1-3), Open-label (Arm 4), Active-comparator (Darbepoetin Alfa) Study of Intermittent Oral Dosing of ASP1517 in Hemodialysis-dependent Chronic Kidney Disease Patients With Anemia
Brief Title: A Study to Investigate the Effect of ASP1517 After Intermittent Oral Dosing in Dialysis Chronic Kidney Disease Patients With Anemia Compared With Darbepoetin as a Reference Drug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1517-CL-0304
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Renal Anemia Associated With Chronic Renal Failure (CRF)
Keywords: Chronic Renal Failure; ASP1517; Renal anemia
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — roxadustat; Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP1517 Low dose group (Experimental): Participants received an oral dose of ASP1517 three times a week.
  Interventions: Drug: roxadustat
- ASP1517 Middle dose group (Experimental): Participants received an oral dose of ASP1517 three times a week.
  Interventions: Drug: roxadustat
- ASP1517 High dose group (Experimental): Participants received an oral dose of ASP1517 three times a week.
  Interventions: Drug: roxadustat
- Darbepoetin group (Active Comparator): Participants received Darbepoetin alfa intravenously once a week.
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: roxadustat — oral
  Other Names: ASP1517
  Arms: ASP1517 High dose group; ASP1517 Low dose group; ASP1517 Middle dose group
Drug: darbepoetin alfa — iv
  Arms: Darbepoetin group

SUMMARY:
This study is to evaluate safety and efficacy of intermittent oral dosing of ASP1517 in dialysis chronic kidney disease patients with anemia.

DETAILED DESCRIPTION:
To evaluate the safety and the dose-response of ASP1517 on hemoglobin (Hb) correction when ASP1517 is applied intermittently in dialysis chronic kidney disease patients with anemia.

To evaluate the treatment effect on Hb maintenance of ASP1517 administered intermittently in dialysis chronic kidney disease patients with anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed as a end-stage kidney disease (ESKD) and are receiving stable chronic maintenance dialysis 3 times per week for ≥ 12 weeks
* Patients who are receiving ESA for at least 8 weeks and the dose of ESA is within the dose range of ESA label
* Hb value at screening test is ≥10.0 g/dL
* Receiving hemodialysis via arteriovenous fistula (AVF) or arteriovenous graft (AVG) or via permanent catheter
* Most recent two Hb values before dialysis during washout period must be both <9.5 g/dL and one of two Hb values must be tested on first visit of the week

Exclusion Criteria:

* Proliferative retinopathy, age-related macular degeneration, retinal vein occlusion and/or macular edema that is considered to require treatment
* Immunological disease with severe inflammation as assessed by the Investigator; even if the inflammation is in remission, the subject is excluded (e.g. lupus erythematosus, rheumatoid arthritis, Sjogren's syndrome, celiac disease, etc)
* Having a history of gastric/intestinal resection considered influential on the absorption of the drug in the gastrointestinal tract or active gastroparesis
* Uncontrollable hypertension (SBP ≥160 mmHg and DBP ≥110 mmHg, before dialysis, at screening test)
* Congestive heart failure (NYHA classification III or higher)
* Having a history of hospitalization for stroke, myocardial infarction or lung infarction within 24 weeks before 1st registration
* Positive for any of the following: human immunodeficiency virus (HIV); hepatitis B surface antigen (HBsAg); or anti-hepatitis C virus antibody (anti-HCV Ab)
* Anemia other than anemia due to low/absent renal production of EPO (e.g., iron deficiency anemia, hemolytic anemia, pancytopenia, etc)
* Pure red cell aplasia
* Using anabolic androgenic steroid, testosterone enanthate or mepitiostane within 6 weeks before 1st registration

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

PRIMARY OUTCOMES:
Rate of rise in hemoglobin (g/dL/week) | Baseline and at Week-6

SECONDARY OUTCOMES:
Cumulative number of responder patients | up to Week-24
  Responder is defined as a hemoglobin >10.0 g/dL and an increase in hemoglobin by >1.0 g/dL from baseline
Percent of visits at which patients maintain hemoglobin between 10.0-12.0 g/dL after achieving hemoglobin ≥10.0 g/dL for each patients | for 28 weeks after dosing
Percent of patients who maintain hemoglobin between 10.0-12.0 g/dL at each visit | for 28 weeks after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokuriku
  - Kansai
  - Kanto
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=355